CLINICAL TRIAL: NCT01187511
Title: Effects of Corticotropin-Releasing Hormone Receptor 1 (CRH1) Antagonism on Stress-Induced Craving in Alcoholic Women With High Anxiety: an Experimental Medicine Study
Brief Title: CRF1 Antagonist GSK561679 in Alcoholism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100046; 10-AA-0046 (Other: NIH)
Record Dates: First submitted 2010-08-21; First posted 2010-08-24 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Alcohol Dependence
Keywords: Addiction; Alcohol Dependence; Anxiety; CRH Antagonist; Stress Induced Craving
MeSH Terms: conditions — Alcoholism; Behavior, Addictive; Anxiety Disorders | interventions — NBI 77860

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK561679 (Active Comparator): GSK561679 was given orally, once a day in the evening, for 21 days, at a dose of 350mg, administered as four tablets consisting of 3 x 100mg tablets plus 1 x 50mg tablet.
  Interventions: Drug: GSK561679
- Placebo (Placebo Comparator): Placebo was given orally, once a day in the evening, for 21 days, in the form of four tablets that matched those of GSK561679
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK561679 — Verucerfont is a corticotropin releasing hormone receptor 1 (CRF1) antagonist.
  Other Names: Verucerfont
  Arms: GSK561679
Drug: Placebo — Placebo is an inactive tablet design to look exactly like GSK561679
  Arms: Placebo

SUMMARY:
Objective:

To evaluate GSK561679, an orally available, brain penetrant selective CRH1 antagonist for its ability to reduce alcohol craving in recently detoxified alcohol dependent women in response to stress or alcohol-associated stimuli.

Study population:

Up to 60 anxious, alcohol dependent women, aged 21-65 years will be enrolled to complete the study in 50 patients.

Background:

* Anxiety, irritability, anger, and depression can all cause stress that may lead to continued drinking in heavy drinkers. One way the brain responds to stress is through a protein on brain cells called a CRH receptor. Previous research has shown that the CRH receptor is involved in negative emotional states and that chronic alcohol consumption increases the activity of CRH receptors in the brain. Medications that block CRH receptors can decrease stress-triggered alcohol consumption.
* GSK561679, an experimental drug that blocks the CRH receptors, can reduce negative emotions such as anxiety and a person s desire for alcohol. By looking at the brain s response to stress and the study drug using functional magnetic resonance imaging (fMRI) scans, researchers hope to learn whether GSK561679 can be an effective treatment for stress-related alcohol abuse.

Objectives:

- To evaluate the usefulness of GSK561679 in reducing stress-related alcohol craving in alcohol-dependent women.

Design:

* Participants in the study will be enrolled in the standard NIH treatment program for alcohol dependence, and will be required to stay at the NIH inpatient treatment unit for an additional 31 days.
* Participants will receive either the study medication or a placebo to be taken once a day in the evening for 4 weeks.
* Participants will have the following procedures while on the study medication:
* Questionnaires about alcohol craving, depression, and anxiety.
* Recordings and responses to personal emotional reactions to stressful, nonstressful, and alcohol-related situations, with blood samples taken during the responses.
* Regular blood tests to measure stress hormones in the blood.
* Speech preparation and presentation (Trier test), along with blood samples, to measure stress hormones in the blood.
* Sessions to measure responses to alcohol-related cues.
* Functional magnetic resonance imaging (fMRI) scans.
* Participants will return for follow-up visits 1 week and 1 month after stopping the study drug and being discharged from the study.

DETAILED DESCRIPTION:
Objective:

To evaluate GSK561679, an orally available, brain penetrant selective CRH1 antagonist for its ability to reduce alcohol craving in recently detoxified alcohol dependent women in response to stress or alcohol-associated stimuli.

Study population:

Up to 60 anxious, alcohol dependent women, aged 21-65 years will be enrolled to complete the study in 50 patients.

Design:

Subjects will be inpatients and enter the present protocol once withdrawal treatment, if needed, is completed. One week of single blind placebo will be followed by randomized double blind treatment with active medication or placebo for approximately 3 weeks. Spontaneous craving for alcohol and ratings of psychopathology will be obtained twice weekly throughout the study. During the placebo lead-in week, a diurnal cortisol curve will be obtained, and a baseline dexamethasone-CRH test may be carried out. These measures will be repeated after 10-14 days of randomized treatment. Around this time, craving responses will also be assessed in a challenge session that combines a social stressor and exposure to physical alcohol cues. During the final week, three sessions of guided imagery will be carried out, on separate days and in a counter-balanced order, exposing the subject to personalized stress-, alcohol- or neutral condition associated stimuli. An fMRI session will be carried out last. Subjects will remain hospitalized throughout the study, and will remain on the unit for a 3 day post-medication monitoring period.

Outcome measures:

The primary outcome will be craving for alcohol on guided imagery challenge sessions. Secondary outcomes will include craving as measured in the combined social stress alcohol cue challenge session, spontaneous craving and psychopathology ratings repeatedly measured on the inpatient unit over time. Exploratory blood biomarkers and brain responses to positive and negative affective stimuli on the fMRI session will also be obtained.

ELIGIBILITY:
* INCLUSION CRITERIA:

DSM-IV diagnosis of alcohol dependence on SCID interview (23), alcohol problems as primary complaint among substance use disorders, and alcohol use within the last month.

Female sex

Spielberger trait anxiety inventory (24) score >39.

Age 21 65 years.

Able to comprehend the consent form, and provide informed consent.

Either:

1. of non-childbearing potential defined as pre-menopausal (for definition, see appendix females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]; or,
2. of child-bearing potential, has a negative serum pregnancy test both on screening and during placebo lead-in, and agrees to one of the following methods of contraception:

i. Practices complete abstinence from intercourse two weeks prior to administration of study drug, throughout participating in the clinical trial and for two weeks following discontinuation of the study medication or,

ii. Has a male sexual partner(s) who is surgically sterilized (vasectomy with documentation of azoospermia) prior to inclusion or,

iii. Has a sexual partner(s) who is/are exclusively female or,

iv. Uses oral contraceptives (either combined or progestogen only) with single-barrier method of contraception consisting of spermicide and condom or diaphragm. Women of child-bearing potential using an oral contraceptive in combination with a single-barrier method of contraception are required to continue to use this form of contraception for 6 weeks following discontinuation of study medication.

v. Uses double-barrier contraception, specifically, a condom plus spermicide and a female diaphragm or cervical cap. The subject must be using this method for at least 2 weeks prior to the administration of the study drug, throughout the study, and 6 weeks following discontinuation of study medication or,

vi. Uses any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year. The subject must have the device inserted at least 2 weeks prior to the first Screen Visit, throughout the study, and 6 weeks following discontinuation of study medication.

EXCLUSION CRITERIA:

1. Investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
2. Employees of GlaxoSmithKline (GSK) or immediate family of GSK employees.
3. Current participation in another clinical study in which the subject is or will be exposed to an investigational or non-investigational drug or device; participation in a clinical study for an illness unrelated to alcohol use within the preceding month; participation in a clinical study related to alcohol use within the preceding six months; or any previous participation in a trial involving GSK561679 or closely related compounds.
4. Inability or unwillingness to participate in an MR scan, including presence of ferromagnetic objects in the body that constitute a contraindication for MRI of the head, or pronounced claustrophobia
5. Any medical or psychiatric condition or laboratory finding other than those explicitly listed below that, in the judgment of the investigator could adversely affect subject safety or study integrity.
6. Schizophrenia, bipolar disease, or any past or present psychotic disorder other than one determined to be substance induced; past or present dementia, or any other disorder which has led to a cognitive impairment that in the opinion of the investigator interferes with the subject s ability to provide informed consent, or comply with study procedures. Any other psychiatric condition which at the present time requires, or in the past month has required pharmacological intervention other than standard withdrawal treatment as described in the NIAAA Assessment and Treatment Protocol.
7. A personality disorder which, in the investigator s judgment could lead to non-compliance with study procedures.
8. Subjects, who in the investigator's judgment, pose a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behavior in the last 6 months and/or any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) (25) in the last 2 months.
9. Unlikely or unable to complete the treatment program because of impending or likely incarceration while on the protocol.
10. Required to receive treatment by a court of law or involuntarily committed to treatment.
11. Positive urine test for illegal drug use.
12. Human Immunodeficiency Virus (HIV) infection.
13. Peptic ulcer disease within the last 10 years, a history of an upper gastro-intestinal (GI) bleeding, or a current stool positive for occult blood (if such stool was obtained without the subject abstaining from red meat for three or more days prior, testing may be repeated once following such abstinence. If that stool is negative for occult blood by the Randomization Day the subject is considered eligible).
14. Any clinically significant liver disease; specifically, cirrhosis as determined by ultrasound; positive test for Hepatitis B surface antigen; positive test for Hepatitis C antibody (hepatitis C antibody positivity confirmed by testing the same sample using a highly specific immunoblot assay, or with hepatitis C RNA test on a separate frozen sample); any of the following liver function test abnormalities:

    1. On screening: gamma glutamyl transpeptidase (GGT) > 5 times the upper limit of normal (ULN), aspartate aminotransferase (AST) > 3 times ULN, alanine transaminase (ALT) > 3 times the ULN or Alkaline Phosphatase > 1.5 ULN; total bilirubin >1.5 times the ULN or direct bilirubin > 35%; Albumin below 3 g/dL; INR > 1.5;
    2. On the day preceding active medication: Alkaline Phosphatase > ULN, AST > 2 times ULN, ALT > 2 times the ULN or GGT > 4 times the ULN, total bilirubin >1.5 times the ULN or direct bilirubin > 35%; Albumin below3 g/dL; INR > 1.5; if, on the day preceding active medication,
    3. On the day preceding active medication, any of the liver function tests above have increased more than 1 time the ULN over the value at the screening.
15. Any cardiovascular condition, including uncontrolled hypertension, or ECG abnormality that, in the investigator s judgment, may pose a safety concern; specifically, ECG finding of a QTc time > 450 msec unless normalized on repeat ECG.
16. Subjects with known or suspected iron deficiency of unknown etiology.
17. Positive pregnancy test, lactating, or planning to become pregnant within 8 weeks from the start of this 4-week study.
18. Regular use of psychotropic medication (antidepressant, lithium, antipsychotic, anxiolytic, antiepileptic, opiates, or hypnotics), within one week, with the exception of benzodiazepines administered within the NIAAA program as part of alcohol withdrawal treatment. Fluoxetine may not have been taken within 5 weeks, and depot antipsychotics may not have been taken within 12 weeks.
19. Current use, or likely requirement during the study, or use of within preceding 4 weeks, of contraindicated medications as listed in Appendix III and 2 weeks for incidental use of non-steroid anti-inflammatory drugs (NSAIDs).
20. Subjects maintained on thyroid medication must have been euthyroid for at least six months.
21. Systemic intake of corticosteroids acutely within two weeks or chronically within the last 6 months (Topical hydrocortisone and inhaled corticosteroids are allowed).
22. A history of allergic reaction to, or significant adverse effects from excipients in the GSK561679 tablet (see GSK561679 Investigator Brochure).

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heilig M, Egli M. Pharmacological treatment of alcohol dependence: target symptoms and target mechanisms. Pharmacol Ther. 2006 Sep;111(3):855-76. doi: 10.1016/j.pharmthera.2006.02.001. Epub 2006 Mar 20. PMID 16545872
- [Background] Heilig M, Koob GF. A key role for corticotropin-releasing factor in alcohol dependence. Trends Neurosci. 2007 Aug;30(8):399-406. doi: 10.1016/j.tins.2007.06.006. Epub 2007 Jul 16. PMID 17629579
- [Background] Epstein DH, Preston KL, Stewart J, Shaham Y. Toward a model of drug relapse: an assessment of the validity of the reinstatement procedure. Psychopharmacology (Berl). 2006 Nov;189(1):1-16. doi: 10.1007/s00213-006-0529-6. Epub 2006 Sep 22. PMID 17019567
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-AA-0046.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK561679 | Placebo
Started | 22 | 22
Completed | 14 | 21
Not Completed | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK561679 | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 21 | 22 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 12 | 17
  White | 16 | 10 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: Alcohol craving was measured using the Alcohol Urges Questionnaire (AUQ). The AUQ is an 8-item self-administered instrument that assesses craving for alcohol among alcohol users in the current context (i.e., right now). The score ranges from 8 (lowest craving value) to 56 (highest craving value).
Time Frame: 15 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 11.6932 (1.6713) | 14.6126 (1.2775)

2. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 15 minutes prior to the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 8.7646 (1.6713) | 10.413 (1.295)

3. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 30 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 11.4075 (1.6713) | 13.0412 (1.2775)

4. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 45 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 9.6218 (1.6713) | 12.1841 (1.2775)

5. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 5 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 13.9789 (1.6713) | 15.946 (1.2775)

6. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 60 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 9.9075 (1.6713) | 12.1841 (1.2775)

7. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 75 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 9.6218 (1.6713) | 11.6603 (1.2775)

8. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 90 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 8.9075 (1.6713) | 13.1841 (1.2775)

9. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 15 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 12.1376 (1.6926) | 13.1086 (1.3065)

10. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 15 minutes prior to the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 9.7805 (1.6926) | 10.6194 (1.297)

11. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 30 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 11.7091 (1.6926) | 13.1432 (1.297)

12. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 45 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 11.3519 (1.6926) | 12.1432 (1.297)

13. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 5 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 14.1376 (1.6926) | 16.9051 (1.297)

14. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 60 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 11.2805 (1.6926) | 12.0956 (1.297)

15. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 75 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 12.2091 (1.6926) | 10.3813 (1.297)

16. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 90 minutes after the beginning of script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 21
Units on a scale | 13.1376 (1.6926) | 10.0004 (1.297)

17. Secondary Outcome: Alcohol Craving in Response to the Trier/Cue-reactivity Procedure
Description: as for outcome 1
Time Frame: 100 minutes after the beginning of the Trier/cue-reactivity procedure, which occurred on Day 21 of the treatment period
Population: The analyses included only those subjects who completed the full Trier/cue-reactivity procedure
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 16 | 21
Units on a scale | 12.977 (2.0207) | 12.0475 (1.7483)

18. Secondary Outcome: Alcohol Craving in Response to the Trier/Cue-reactivity Procedure
Description: as for outcome 1
Time Frame: 15 minutes prior to the beginning of the Trier/cue-reactivity procedure, which occurred on Day 21 of the treatment period
Population: The analyses included only those subjects who completed the full Trier/cue-reactivity procedure
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 16 | 21
Units on a scale | 15.1645 (2.0207) | 12.0116 (1.7163)

19. Secondary Outcome: Alcohol Craving in Response to the Trier/Cue-reactivity Procedure
Description: as for outcome 1
Time Frame: 20 minutes after the beginning of the Trier/cue-reactivity procedure, which occurred on Day 21 of the treatment period
Population: The analyses included only those subjects who completed the full Trier/cue-reactivity procedure
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 16 | 21
Units on a scale | 18.4145 (2.0207) | 15.2497 (1.7163)

20. Secondary Outcome: Alcohol Craving in Response to the Trier/Cue-reactivity Procedure
Description: as for outcome 1
Time Frame: 40 minutes after the beginning of the Trier/cue-reactivity procedure, which occurred on Day 21 of the treatment period
Population: The analyses included only those subjects who completed the full Trier/cue-reactivity procedure
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 16 | 21
Units on a scale | 20.352 (2.0207) | 18.0116 (1.7163)

21. Secondary Outcome: Alcohol Craving in Response to the Trier/Cue-reactivity Procedure
Description: as for outcome 1
Time Frame: 70 minutes after the beginning of the Trier/cue-reactivity procedure, which occurred on Day 21 of the treatment period
Population: The analyses included only those subjects who completed the full Trier/cue-reactivity procedure
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 16 | 21
Units on a scale | 13.7895 (2.0207) | 13.0592 (1.7163)

22. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: Anxiety symptoms were measured using the Comprehensive Psychopathological Rating Scale (CPRS). The CPRS is an 18-item interview-based instrument for assessing depression and anxiety. There are two 10-item subscales, the Montgomery-Asberg Depression Rating Scale (MADRS) and the Brief Scale for Anxiety (BSA). Each subscale ranges from 0 (lowest symptom severity) to 60 (highest symptom severity).
Time Frame: Day 1 of the treatment period
Population: The analyses included only those subjects who had a baseline anxiety symptom rating taken 1 day after inpatient admission (but prior to enrollment in this protocol), and who completed all 32 days of the treatment period
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 7.8582 (1.2811) | 8.7076 (1.0221)

23. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 22
Time Frame: Day 11 of the treatment period
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 6.4777 (1.2117) | 7.041 (1.0221)

24. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 22
Time Frame: Day 14 of the treatment period
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 6.5443 (1.2117) | 6.6122 (1.0558)

25. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 22
Time Frame: Day 18 of the treatment period
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 6.011 (1.2117) | 5.4219 (1.0221)

26. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 22
Time Frame: Day 21 of the treatment period
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 6.611 (1.2117) | 5.7835 (1.0386)

27. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 22
Time Frame: Day 25 of the treatment period
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 5.3112 (1.239) | 5.1362 (1.0221)

28. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 22
Time Frame: Day 28 of the treatment period
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 7.2231 (1.2449) | 4.5648 (1.0221)

29. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 22
Time Frame: Day 32 of the treatment period
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 5.2365 (1.2878) | 4.2791 (1.0221)

30. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 22
Time Frame: Day 4 of the treatment period
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 6.6777 (1.2117) | 5.9457 (1.0221)

31. Secondary Outcome: Anxiety Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 22
Time Frame: Day 7 of the treatment period
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 6.6078 (1.2379) | 6.66 (1.0221)

32. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: Depression symptoms were measured using the Comprehensive Psychopathological Rating Scale (CPRS). The CPRS is an 18-item interview-based instrument for assessing depression and anxiety. There are two 10-item subscales, the Montgomery-Asberg Depression Rating Scale (MADRS) and the Brief Scale for Anxiety (BSA). Each subscale ranges from 0 (lowest symptom severity) to 60 (highest symptom severity).
Time Frame: Day 1 of the treatment period
Population: The analyses included only those subjects who had a baseline depression symptom rating taken 1 day after inpatient admission (but prior to enrollment in this protocol), and who completed all 32 days of the treatment period
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 10.002 (1.4252) | 8.7759 (1.1)

33. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 32
Time Frame: Day 11 of the treatment period
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 6.3187 (1.3626) | 6.2997 (1.1)

34. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 32
Time Frame: Day 14 of the treatment period
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 7.6521 (1.3626) | 8.0633 (1.1268)

35. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 32
Time Frame: Day 18 of the treatment period
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 8.0521 (1.3626) | 6.5855 (1.1)

36. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 32
Time Frame: Day 21 of the treatment period
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 7.0521 (1.3626) | 5.9353 (1.1142)

37. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 32
Time Frame: Day 25 of the treatment period
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 4.8092 (1.3845) | 4.9188 (1.1)

38. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 32
Time Frame: Day 28 of the treatment period
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 7.149 (1.3958) | 4.2997 (1.1)

39. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 32
Time Frame: Day 32 of the treatment period
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 4.8071 (1.4396) | 4.2045 (1.1)

40. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 32
Time Frame: Day 4 of the treatment period
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 8.2521 (1.3626) | 7.1569 (1.1)

41. Secondary Outcome: Depression Symptom Ratings Measured Bi-weekly During the Treatment Period
Description: as for outcome 32
Time Frame: Day 7 of the treatment period
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 6.6366 (1.383) | 6.9188 (1.1)

42. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: Alcohol craving was measured using the Penn Alcohol Craving Scale (PACS). The PACS is a five-item self-administered instrument for assessing alcohol craving over the course of the past week. The score ranges from 0 (lowest craving value) to 30 (highest craving value).
Time Frame: Day 1 of the treatment period
Population: The analyses included only those subjects who had a baseline craving measure taken 4 days after inpatient admission (but prior to enrollment in this protocol), and who completed all 32 days of the treatment period
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 9.5572 (1.4164) | 12.2152 (1.1474)

43. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 42
Time Frame: Day 11 of the treatment period
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 7.7 (1.4164) | 8.8468 (1.1474)

44. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 42
Time Frame: Day 14 of the treatment period
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 5.7 (1.4164) | 7.3205 (1.1474)

45. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 42
Time Frame: Day 18 of the treatment period
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 6.2715 (1.4164) | 6.9521 (1.1474)

46. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 42
Time Frame: Day 21 of the treatment period
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 5.2715 (1.4164) | 6.531 (1.1474)

47. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 42
Time Frame: Day 25 of the treatment period
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 4.6286 (1.4164) | 6.6363 (1.1474)

48. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 42
Time Frame: Day 28 of the treatment period
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 3.6083 (1.4455) | 6.5836 (1.1474)

49. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 42
Time Frame: Day 32 of the treatment period
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 3.7666 (1.4634) | 6.531 (1.1474)

50. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 42
Time Frame: Day 4 of the treatment period
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 7.9858 (1.4164) | 9.7942 (1.1474)

51. Secondary Outcome: Spontaneous Alcohol Craving Measured Bi-weekly During the Treatment Period
Description: as for outcome 42
Time Frame: Day 7 of the treatment period
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 14 | 19
Units on a scale | 8.1286 (1.4164) | 8.7942 (1.1474)

ADVERSE EVENTS:
Arm/Group | GSK561679 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 22/22 | 22/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK561679 (N=22) | Placebo (N=22)
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 7 | 7
Heartburn (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 9 | 7
Stomach pain (Gastrointestinal disorders) | 7 | 10
Upset Stomach (Gastrointestinal disorders) | 8 | 8
Fatigue (General disorders) | 15 | 15
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Dizziness (Nervous system disorders) | 9 | 5
Headache (Nervous system disorders) | 19 | 15
Somnolence (Nervous system disorders) | 21 | 20
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 15 | 12
Acne (Skin and subcutaneous tissue disorders) | 11 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No